CLINICAL TRIAL: NCT05753800
Title: Efficacy of the INTORUS Device as a Therapeutic Tool in Motor Intervention
Brief Title: Efficacy of INTORUS as a Therapeutic Tool in Motor Intervention in Patients at Aspace Centres in the Province of Cáceres
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Extremadura (Other)
Responsible Party: Principal Investigator, Blanca González Sanchez, doctor, University of Extremadura
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IPC.2023
Record Dates: First submitted 2023-01-30; First posted 2023-03-03 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Cerebral Palsy; Motor Disorders; Motor Activity
Keywords: cerebral palsy; motor activity; motor disorders
MeSH Terms: conditions — Cerebral Palsy; Motor Disorders; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): This group receives motor intervention sessions with the Intorus device
  Interventions: Device: INTORUS
- Control group (No Intervention): This group receives no motor intervention sessions with the Intorus device

INTERVENTIONS:
Device: INTORUS — Motor intervention protocol with Intorus consisting of a series of exercises of progressive difficulty
  Arms: Experimental group

SUMMARY:
The goal of this Clinical Trial is to verify the effectiveness of the use of the Intorus device in the motor intervention in patients with cerebral palsy and related syndromes. The main question it aims to answer is:

Does the use of the Intorus tool manage to improve the mobility of upper limbs (MMSS) in patients with infantile cerebral palsy to increase their performance in activities of daily living? A total of approximately 50 users will participate in the study. Participants will be divided into two groups randomly. The control group will receive an intervention treatment at the motor level in the traditional way, following the protocols established in the center, and the intervention group will receive an intervention treatment at the motor level with the INTORUS device.

Randomization will be carried out using the Oxford Minimization and Randomization software.

DETAILED DESCRIPTION:
The intervention program will take place during the Occupational Therapy sessions and will be carried out by the center's occupational therapists. These sessions must be carried out in a quiet environment, without distractions so that the user can concentrate on carrying out the activities. It is important that the patient attends the sessions in comfortable, sleeveless clothing, to allow the tool to slide smoothly through their upper limbs.

Each session will consist of several exercises with their corresponding rest breaks.

EVALUATION

The evaluations will be carried out prior to the start of treatment, at 20 weeks of treatment and at 40 weeks of treatment once the intervention program has concluded.

The tools used to carry out the evaluation will be:

* Questionnaire of sociodemographic variables
* Goniometric

  * Shoulder joint: abduction-adduction, flexion-extension, external-internal rotation.
  * Elbow joint: flexion-extension, pronation-supination.
  * Wrist joint: flexion-extension, radial-ulnar deviation.
  * Articulation of the thumb: abduction-adduction, flexion-extension, opposition.
  * Articulation of the fingers: flexion-extension, abduction-adduction.
* Gross Motor Function Classification
* Assessment of a functional gesture
* Satisfaction questionnaire for professionals The evaluations will be carried out by a professional external to the center to avoid bias.

Once the intervention period is over, a questionnaire will be passed to the professionals participating in the study to assess the usefulness of the device, the degree of satisfaction with it and the usefulness of the therapies applied.

TIMELINE The intervention consists of 40 treatment sessions lasting 45 minutes each with a frequency of 2 days a week in which the intervention program described above will be developed.

Previously, the participants will receive a "session 0" in which they will carry out a first contact with the device.

ELIGIBILITY:
Inclusion Criteria:

* Users with infantile cerebral palsy and/or related syndromes.
* Ages between 4 and 18 years.
* Motor disability.
* Affectation in the mobility of upper limbs.
* Informed consent signed by parents/guardians.

Exclusion Criteria:

* Patients with another type of pathology not related to cerebral palsy.
* Under 4 years and over 18 years.
* Participants who do not meet the inclusion criteria described above

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
IMPROVEMENT OF UPPER LIMB MOBILITY AS MEASURED BY GONIOMETER | Before starting treatment. After 20 weeks of treatment and at the end of treatment (40 weeks).
  Measuring joint amplitude of upper limb joints with goniometer

SECONDARY OUTCOMES:
Functional Gesture of Activities of Daily Living | Before starting treatment. After 20 weeks of treatment and at the end of treatment (40 weeks).
  Measurement of the performance of a functional gesture performed in the patient's activities of daily living.

OTHER OUTCOMES:
Professional satisfaction questionnaire | Through study completion, an average of 6 months
  Measurement of professionals' satisfaction with the use of the tool measured with a questionnaire designed by ourselves.
Participants satisfaction questionnaire | Through study completion, an average of 6 months
  Measurement of participants' satisfaction with the use of the tool measured with a questionnaire designed by us.

CONTACTS AND LOCATIONS:
Overall Officials: Blanca González Sánchez, Doctor, Principal Investigator — Universidad de Extremadura
Locations (1):
- Blanca González Sánchez, Cáceres, Caceres, Spain

IPD SHARING:
Plan to Share IPD: No